CLINICAL TRIAL: NCT02982564
Title: Effect of Low-intensity Versus Moderate-intensity Endurance Exercise on Physical Functioning Among Breast Cancer Survivors: a Randomized Controlled Trial
Brief Title: Effect of Low vs Moderate-intensity Endurance Exercise on Physical Functioning Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1SC3GM116684-01 (NIH)
Record Dates: First submitted 2016-11-23; First posted 2016-12-05 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Breast Neoplasms
Keywords: Exercise; Physical Functioning; Hispanic
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Intensity Exercise (Experimental): Participants engage in low intensity endurance exercise.
  Interventions: Behavioral: Exercise Program Low Intensity
- Moderate Intensity Exercise (Experimental): Participants engage in moderate intensity endurance exercise.
  Interventions: Behavioral: Exercise Program Moderate Intensity

INTERVENTIONS:
Behavioral: Exercise Program Low Intensity — This arm includes a low-intensity intervention and will have a duration of six months. Participants will be provided with a heart rate monitor to train at the intensity according to group assignment. Progression for both programs in the endurance component will be slower and more gradual for deconditioned participants, and may require multiple shorter periods (5-10 minutes) with rest intervals.
  Arms: Low Intensity Exercise
Behavioral: Exercise Program Moderate Intensity — This arm includes a moderate-intensity intervention and will have a duration of six months. Participants will be provided with a heart rate monitor to train at the intensity according to group assignment. Progression for both programs in the endurance component will be slower and more gradual for deconditioned participants, and may require multiple shorter periods (5-10 minutes) with rest intervals.
  Arms: Moderate Intensity Exercise

SUMMARY:
The purpose of this study is to evaluate the effect of two exercise programs: 1) one program will be at low intensity; 2) the other program will be at moderate intensity. One hundred forty two women who are breast cancer survivors will be recruited. Participants will be educated on a home exercise program to be performed at either low or moderate intensity, according to group assignment. Evaluations to participants will consist of function and quality of life.

DETAILED DESCRIPTION:
Improvements in early diagnosis and treatment for breast cancer in women have resulted in increased survivorship. An unintended consequence of increased survival, however, is that more women are living with the negative sequelae associated with cancer treatment, including decreased physical function. Exercise has been beneficial in arresting these sequelae, but adherence to exercise guidelines continues to be a challenge. As most breast cancer survivors are middle-aged and older, an alternative to enhance exercise engagement and adherence might be providing a low intensity exercise program. The overall purpose of this study is to assess the impact of a low intensity versus moderate intensity endurance exercise program on physical functioning on breast cancer survivors. It is hypothesized that participants of the low intensity exercise program will demonstrate similar physical functioning as participants in the moderate intensity exercise program. The Theory of Planned Behavior will serve as framework for the intervention. A convenience sample of 142 women, residents of Puerto Rico, age 50 or older, with a diagnosis of breast cancer, stage 0 thru III, who have received surgical treatment for breast cancer, with or without adjuvant therapy, will be randomly assigned to a low intensity or moderate intensity endurance intervention. Both interventions will be home-based, have a duration of 6 months, and be provided by physical therapists. An evaluator blinded to group assignment will assess participants at baseline and at completion of the intervention. Primary outcome measures will consist of physical functioning, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Fifty years of age or older
2. Be a resident of the San Juan metropolitan area of Puerto Rico (PR)
3. Diagnosed with breast cancer
4. Be classified in breast cancer stage grouping 0 to III according to the American Joint Committee on Cancer Classification of Malignant Tumors (TNM) Staging System (2013)
5. Have completed adjuvant curative therapy at least two months to 5 years prior to recruitment

Exclusion Criteria:

1. Women who have contraindications to exercise, such as extreme fatigue or anemia, unstable cardiac disease; uncontrolled diabetes; uncontrolled hypertension; coagulopathies; inability to ambulate independently
2. Women with metastasis or secondary cancers
3. Women who already meet the national standard for exercise (≥ 150 minutes per week of moderate exercise).

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Change in Cardiovascular fitness: Six-minute walk test | At month 1 prior to intervention (pre-test); at 6-month (post-test); 6-month follow up.
  Will be used to assess physical function in cancer survivors. It has been validated to assess exercise tolerance (American Thoracic Society, 2002) and has been recommended as a test suitable for fitness, as it is highly correlated with oxygen uptake. An increase in walking distance indicates an improvement in performance. Data will be collected on distance walked (meters), number of rests, and duration of rest during the 6 minutes. Rating of perceived exertion will be monitored. Heart rate and oxygen saturation will be examined using a pulse oximeter.
Change in Quality of Life | At month 1 prior to intervention (pre-test); at 6-month (post-test); 6-month follow up.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v.1.0/1.1 General Health. The Spanish version (Salud general) will be used. It contains two subdomains: Global Physical Health and Global Mental Health. The final score can be converted to a score for the EUROQoL.
Change in Functioning | At month 1 prior to intervention (pre-test); at 6-month (post-test); 6-month follow up.
  PROMIS Item Bank v. 1.2 Physical Function. The Spanish version (Capacidad de Funcionamiento Físico - Cuestionario Abreviado 20) will be used. It consists of 20 items, measuring upper extremity function, as well as gross motor function such as walking and stairs use.
Change in Depression | At month 1 prior to intervention (pre-test); at 6-month (post-test); 6-month follow up.
  Inventario -II de depresión de Beck (BDI-II). The Spanish version has proper psychometric properties for assessment of depression (internal consistency, obtaining a Cronbach alfa of 0.89 and has reported known-group validity; Vega-Dienstmaier, 2014).
Change in Body Image | At month 1 prior to intervention (pre-test); at 6-month (post-test); 6-month follow up.
  Body Appreciation Scale-2 (BAS-2; Tylka & Wood-Barcalow, 2014), Spanish version will be used to measure body appreciation, an aspect that encompasses positive self-evaluation of body image. It has 13 items with responses ranging from 1 (never) to 5 (always). The Spanish BAS showed adequate internal consistency (Cronbach's α = .91) and construct validity (correlations with BMI, influence of the body shape model, perceived stress, coping strategies, self-esteem and variables from the Eating Disorders Inventory-2). Test-retest reliability ranged from .88 to .90.

SECONDARY OUTCOMES:
Change in Physical Activity | At month 1 prior to intervention (pre-test); at 6-month (post-test); 6-month follow up.
  Accelerometers will be used to evaluate the amount of time spent in low to moderate and moderate to vigorous physical activity. Accelerometry has been found to be a valid measure of physical activity, as compared to oxygen uptake and calorimetry (Hendelman et al., 2000; Kuffel, et al., 2011) and has been used nationally by the National Health and Nutritional Examination Survey (NHANES) study to document, more precisely than self-reported measures, the intensity and time of physical activity (Hawkins et al., 2009). The procedures established by NHANES (CDC, 2005) will be followed.
Change in Time spend in Habitual Physical Activities | At month 1 prior to intervention (pre-test); at 6-month (post-test); 6-month follow up.
  International Physical Activity Questionnaire (IPAQ, 2002, self-administered, long Spanish version). The IPAQ assesses multiple domains of activity such as leisure, occupation, household, and transport, among others (Craig et al., 2003). This questionnaire has proved to be reliable (Roman-Viñas et al., 2010), and has been validated with accelerometer, pedometer, physical activity log, and maximal oxygen uptake (van Poppel et al., 2010).
Adherence | At 6-month follow up.
  Exercise logs. Participants will be asked to record week number and type and duration of exercise. Logs will be collected at the 6-month evaluation session.

CONTACTS AND LOCATIONS:
Overall Officials: Ana L Mulero-Portela, PhD, Principal Investigator — University of Puerto Rico Medical Sciences Campus
Locations (1):
- Puerto Rico Clinical and Translational Research Consortium, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Data will be presented at the conclusion of the study.

REFERENCES:
- [Derived] Mulero Portela AL, Colon Santaella CL, Rogers LQ, Missaghian Vissepo M. Effect of low- and moderate-intensity endurance exercise on physical functioning among breast cancer survivors: a randomized controlled trial. Support Care Cancer. 2024 Dec 21;33(1):49. doi: 10.1007/s00520-024-09100-2. PMID 39714637